CLINICAL TRIAL: NCT00381992
Title: Risk Assessment of Long-Haul Truck Drivers
Status: Completed | Type: Observational
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH); University of Alabama at Birmingham (Other)
Responsible Party: Sponsor
Other Study IDs: F060815005; 5R34MH073411-03 (NIH)
Record Dates: First submitted 2006-09-26; First posted 2006-09-28 (Estimated); Last update posted 2017-11-07 (Actual); Status verified 2014-12

CONDITIONS: Gonorrhea; Chlamydia Infections; Hepatitis B; Hepatitis C; Diabetes Mellitus; Hypertension; Obesity; HIV Infections; Hyperlipidemia
Keywords: sexual risk behavior; diabetes mellitus; hypertension; obesity; human immunodeficiency virus; hyperlipidemia; chlamydia
MeSH Terms: conditions — Gonorrhea; Chlamydia Infections; Hepatitis B; Hepatitis C; Diabetes Mellitus; Hypertension; Obesity; HIV Infections; Hyperlipidemias; Acquired Immunodeficiency Syndrome

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

SUMMARY:
International studies have repeatedly documented a substantial prevalence of sexual risk behaviors and high rates of human immunodeficiency virus (HIV) and other sexually transmitted infections (STI) ranging from 5%-56% amongst long-distance truck drivers ("truckers") living in diverse international settings including India, Bangladesh, South Africa, China, Laos and Thailand. The prevalence of sexual risk factors and STI/HIV in US drivers is unknown. This proposal will provide both qualitative and quantitative data on HIV risk behaviors by interviewing and testing truckers working for established long-distance trucking firms, the sector which accounts for most of the jobs in the trucking and warehousing industry in the United States. The data obtained from this study will be used to inform the development of an HIV prevention intervention for long-haul truck drivers.

DETAILED DESCRIPTION:
The study proposed in this R34 application will address the following specific aims:

Specific Aim 1. To perform focus groups and in-depth interviews with long-haul truck drivers to guide development of both a behavioral risk assessment instrument and an acceptable HIV/STI screening protocol for long-haul truckers.

Specific Aim 2. To perform in-depth interviews with trucking industry executives to determine barriers to routine HIV/STI assessment and screening of their employees.

Specific Aim 3. To perform a pilot phase with a subsample of long-haul truck drivers characterized by the following steps: TTM-based "cognitive interviews" (N=5); pilot testing of the survey and biomedical screening protocol (N=15); and a follow-up focus group (N=8)

Specific Aim 4. To assess a sample of (N=300) truck drivers for general health and sexual risk behaviors using the adapted theory-based survey and to determine the prevalence of hepatitis B, hepatitis C, hypertension, hyperlipidemia, diabetes and obesity, HIV, N. gonorrhoeae, and C. trachomatis

ELIGIBILITY:
Inclusion Criteria:

1. Long-haul truck driver as defined as a driver, part-time or full-time, who drives a truck across state lines (interstate)
2. English speaking
3. Age 21 or greater
4. Willing to participate
5. Able to provide written informed consent

Exclusion Criteria:

1. Does not fit definition of truck driver in inclusion criteria #1
2. Unwilling to participate
3. Unwilling or unable to provide informed consent
4. Unable to understand or speak English
5. Age < 21 years

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: American long-haul truck drivers affiliated with participating companies or presenting as clients at participating truck stops.
Sampling Method: Non-Probability Sample
Enrollment: 294 (Actual)
Dates: Start 2005-09; Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

PRIMARY OUTCOMES:
The prevalence of hepatitis B, hepatitis C, hypertension, hyperlipidemia, diabetes and obesity, HIV, N. gonorrhoeae, and C. trachomatis | Cross-sectional

CONTACTS AND LOCATIONS:
Overall Officials: Laura H Bachmann, MD, MPH, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Wake Forest University Health Sciences, Winston-Salem, North Carolina, United States

REFERENCES:
- [Result] Lichtenstein B, Hook EW 3rd, Grimley DM, St Lawrence JS, Bachmann LH. HIV risk among long-haul truckers in the USA. Cult Health Sex. 2008 Jan;10(1):43-56. doi: 10.1080/13691050701582936. PMID 18038280